CLINICAL TRIAL: NCT03450486
Title: Effects of Exercise on Joint Stiffness and Dynamic Balance in Individuals With Knee Osteoarthritis Evaluated Through Star Excursion Balance Test
Brief Title: Exercise on Knee OA With the Star Excursion Balance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 110819
Record Dates: First submitted 2018-02-20; First posted 2018-03-01 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
Keywords: dynamic balance; star excursion balance test; exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will include one intervention arm and one control arm. The intervention arm will include balance measurements from the affected side of individuals with unilateral knee osteoarthritis. The control arm will will include balance measurements from the unaffected side of individuals with unilateral knee osteoarthritis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- affected limb (Experimental): measurements of balance from the affected side of individuals with unilateral knee osteoarthritis following an exercise session
  Interventions: Other: exercise
- unaffected limb (Active Comparator): measurements of balance from the unaffected side of individuals with unilateral knee osteoarthritis following an exercise session
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — one 30 minute bout of mild exercise

SUMMARY:
Osteoarthritis is a prevalent and disabling condition. Exercise is recommended to maintain strength and mobility, and to decrease pain. However, acute bouts of exercise have conflicting outcomes: they are fatiguing and they also can increase coordination and balance. The purpose of this study is to assess the effects of a single bout of exercise (30 minutes) on balance performance of individuals with self-identified unilateral knee osteoarthritis. Balance will be assessed using the star excursion balance test before and after the exercise session. Differences in performance between the two star excursion balance tests will reflect the changes due to exercise. The changes between their balance performance on each limb will reflect the changes due to osteoarthritis.

DETAILED DESCRIPTION:
Knee OA affects over 241 million people worldwide, and poses a significant burden to the healthcare system (Cross et al., 2014). Knee OA leads to decreased quadriceps muscle strength, and impaired postural control and joint proprioception (Hurley et al., 1997). These factors lead to balance impairments in individuals with osteoarthritis compared to controls (Wegener et al., 1997). It has been reported that the completion of a warm-up program improves the dynamic and static balance of healthy individuals (Daneshjoo et al., 2012). Therefore, exercise may acutely facilitate neuromuscular control, reduce stiffness and significantly improve dynamic balance in individuals with knee OA. Alternatively, muscular fatigue that may negate these benefits (Nardone et al., 1997). Given that falls are a devastating injury in the elderly (Sri-On et al, 2017), and that exercise programs improve balance (Carter et al, 2001; Tse et al, 2015) it is important to evaluate the acute effects of a single bout of exercise on balance performance in individuals with osteoarthritis. The Star Excursion Balance Test (SEBT) has been validated for quantifying dynamic balance in healthy individuals (Kinzey & Armstrong, 1998) and individuals with knee OA (Kanko, 2017). It is important to evaluate the effects of exercise on balance in individuals with OA as changes in balance following exercise may lead to either impairments or improvements, and have direct implications for the safety of exercise as a recommended approach in OA.

This study will recruit 35 individuals with self-identified unilateral knee osteoarthritis, according to clinical criteria for classification of idiopathic knee OA (Altman et al., 1986). They will complete a Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) to clear them for participation in physical activity (Warburton et al, 2011). They will complete a standard questionnaire assessing knee function: the Knee injury and Osteoarthritis Outcome Score (KOOS) (Roos et al, 2003). They will complete the star excursion balance test, on each of their affected and unaffected limbs, before and after completing a 30 minute bout of exercise. This exercise session will be supervised, and emphasizes optimal alignment of the trunk and lower limb joints relative to one another, as well as quality of movement performance, while dynamically and functionally strengthening the lower limb muscles (Bennell et al, 2011). The research participants will dictate the intensity and duration of the program.

Differences in performance between the two star excursion balance tests will reflect the changes due to exercise. The changes between their balance performance on each limb will reflect the changes due to osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* unilateral knee osteoarthritis according to clinical criteria for classification of idiopathic osteoarthritis (OA) of the knee (Altman et al., 1986)
* routinely engaging in mild exercise, such as walking or gardening.
* a completed PAR-Q+ indicating no contraindications

Exclusion Criteria:

* lower extremity joint replacement
* Inflammatory or Infectious Arthritis
* Major neurological disorder (ex. Parkinson's disease, Huntington's disease, Multiple Sclerosis, peripheral neuropathy)
* Major medical illness that would interfere with participating in a 30 minute bout of exercise
* Inability to engage in moderate physical activity for 30-40 minutes
* Inability to read English
* Psychiatric illness that limits informed consent
* Inability to stand on limb for more than 5 seconds

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
star excursion balance test | change in star excursion balance test after the 30 minute bout of exercise
  standard test for assessing dynamic balance. Individuals stand on one limb and reach their other limb in each of eight directions (eg anterior, lateral, antero-lateral, etc) and the length of the reach is measured. The reach measurements are normalized by dividing by leg length.

CONTACTS AND LOCATIONS:
Overall Officials: James P Dickey, PhD, Principal Investigator — Western University
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Each participant will be identified with a code (eg. STAR001) that correlates to his or her addition to the study. The master sheet will be the only document that contains the decoding system, and will be stored in a locked filing cabinet. All other data will be labeled using the participant's identification code.

REFERENCES:
- [Background] Roddy E, Zhang W, Doherty M, Arden NK, Barlow J, Birrell F, Carr A, Chakravarty K, Dickson J, Hay E, Hosie G, Hurley M, Jordan KM, McCarthy C, McMurdo M, Mockett S, O'Reilly S, Peat G, Pendleton A, Richards S. Evidence-based recommendations for the role of exercise in the management of osteoarthritis of the hip or knee--the MOVE consensus. Rheumatology (Oxford). 2005 Jan;44(1):67-73. doi: 10.1093/rheumatology/keh399. Epub 2004 Sep 7. PMID 15353613
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Hurley MV, Scott DL, Rees J, Newham DJ. Sensorimotor changes and functional performance in patients with knee osteoarthritis. Ann Rheum Dis. 1997 Nov;56(11):641-8. doi: 10.1136/ard.56.11.641. PMID 9462165
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Wegener L, Kisner C, Nichols D. Static and dynamic balance responses in persons with bilateral knee osteoarthritis. J Orthop Sports Phys Ther. 1997 Jan;25(1):13-8. doi: 10.2519/jospt.1997.25.1.13. PMID 8979171
- [Background] Daneshjoo A, Mokhtar AH, Rahnama N, Yusof A. The effects of comprehensive warm-up programs on proprioception, static and dynamic balance on male soccer players. PLoS One. 2012;7(12):e51568. doi: 10.1371/journal.pone.0051568. Epub 2012 Dec 12. PMID 23251579
- [Background] Nardone A, Tarantola J, Giordano A, Schieppati M. Fatigue effects on body balance. Electroencephalogr Clin Neurophysiol. 1997 Aug;105(4):309-20. doi: 10.1016/s0924-980x(97)00040-4. PMID 9284239
- [Background] Sri-On J, Tirrell GP, Bean JF, Lipsitz LA, Liu SW. Revisit, Subsequent Hospitalization, Recurrent Fall, and Death Within 6 Months After a Fall Among Elderly Emergency Department Patients. Ann Emerg Med. 2017 Oct;70(4):516-521.e2. doi: 10.1016/j.annemergmed.2017.05.023. Epub 2017 Jul 5. PMID 28688769
- [Background] Carter ND, Kannus P, Khan KM. Exercise in the prevention of falls in older people: a systematic literature review examining the rationale and the evidence. Sports Med. 2001;31(6):427-38. doi: 10.2165/00007256-200131060-00003. PMID 11394562
- [Background] Tse AC, Wong TW, Lee PH. Effect of Low-intensity Exercise on Physical and Cognitive Health in Older Adults: a Systematic Review. Sports Med Open. 2015;1(1):37. doi: 10.1186/s40798-015-0034-8. Epub 2015 Oct 20. PMID 26512340
- [Background] Kinzey SJ, Armstrong CW. The reliability of the star-excursion test in assessing dynamic balance. J Orthop Sports Phys Ther. 1998 May;27(5):356-60. doi: 10.2519/jospt.1998.27.5.356. PMID 9580895
- [Background] Bennell KL, Egerton T, Wrigley TV, Hodges PW, Hunt M, Roos EM, Kyriakides M, Metcalf B, Forbes A, Ageberg E, Hinman RS. Comparison of neuromuscular and quadriceps strengthening exercise in the treatment of varus malaligned knees with medial knee osteoarthritis: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2011 Dec 5;12:276. doi: 10.1186/1471-2474-12-276. PMID 22141334
- [Background] Kanko L:
- [Background] Warburton DE, Gledhill N, Jamnik VK, Bredin SS, McKenzie DC, Stone J, Charlesworth S, Shephard RJ. Evidence-based risk assessment and recommendations for physical activity clearance: Consensus Document 2011. Appl Physiol Nutr Metab. 2011 Jul;36 Suppl 1:S266-98. doi: 10.1139/h11-062. PMID 21800945